CLINICAL TRIAL: NCT04897659
Title: Persistent Left Bundle Branch Block After Rapid-Deployment Aortic Valve Replacement: Incidence, Long-term Prognostic and Predictive Factors
Brief Title: Left Bundle Branch Block (LBBB) After IntuityTM
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: CIL 2019-48 bis
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate incidence, prognosis and predictive factors of new-onset of persistent left bundle branch block (LBBB) after rapid-deployment aortic valve replacement (RD-AVR) with the IntuityTM bioprosthesis.

It was an observational, retrospective and single-center study. Two hundred and seventy-four consecutive patients without any baseline ventricular conduction disorder or previous permanent pacemaker or defibrillator implantation who underwent RD-AVR with the IntuityTM valve were included. Twelve-lead electrocardiogram and transthoracic echocardiography were performed preoperatively, postoperatively, at discharge, 1-month, and 1-year. Incidence, prognosis and predictive factors of new-onset of persistent LBBB were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* rapid-deployment aortic valve replacement (RD-AVR) with the Edwards Intuity™ bioprosthesis for severe aortic valve stenosis
* between July 2012 and May 2018

Exclusion Criteria:

* preoperative permanent pacemaker or defibrillator,
* complete intraventricular conductive disorder defined by a QRS width ≥ 120 ms.
* absence of patient's authorization for anonymous publication of their clinical data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred and seventy-four consecutive patients without any baseline ventricular conduction disorder or previous permanent pacemaker or defibrillator implantation who underwent rapid-deployment aortic valve replacement (RD-AVR) with the IntuityTM valve were included. Twelve-lead electrocardiogram and transthoracic echocardiography were performed preoperatively, postoperatively, at discharge, 1-month, and 1-year.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of NOP-LBBB (new onset of persistent left bundle branch block) | at 1 year
  QRS duration ≥ 120 ms with QS or rS patterns on the V1 lead, a large notched R wave in D1, aVL, V5 and V6 and the absence of Q wave in V5 and V6, according to the recommendations of the American Heart Association. NOP-LBBB was persistence of LBBB on the 12-lead recording electrocardiogram (ECG) at discharge from hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France